CLINICAL TRIAL: NCT01983371
Title: Diagnostic Accuracy of Ferumoxytol-Enhanced MRI for Detecting Lymph Node Metastases in Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Scott Potenta, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Scott Potenta, MD, PhD, Clinical Instructor, University of Vermont
Organization: University of Vermont (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRMS 14-096
Record Dates: First submitted 2013-11-05; First posted 2013-11-14 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferumoxytol-enhanced MRI (Experimental): This is a single-arm study. All enrolled patients will have a ferumoxytol-enhanced MRI scan.
  Interventions: Drug: Ferumoxytol; Other: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol — All study patients will receive a dose of ferumoxytol for the MRI. Ferumoxytol will be administered intravenously at a dose of 6 mg/kg, for a maximum dose of 510 mg.
  Other Names: Feraheme
Other: Magnetic Resonance Imaging — All study patients will undergo a ferumoxytol-enhanced MRI in addition to any other ongoing care for colorectal cancer. Histopathologic analysis of lymph nodes will be the gold standard for determining lymph node status.
  Other Names: MRI

SUMMARY:
The purpose of this study is to determine the diagnostic accuracy of ferumoxytol-enhanced MRI in detecting lymph nodes that have been invaded by tumor cells in patients with colorectal cancer.

DETAILED DESCRIPTION:
This study will investigate the accuracy of ferumoxytol-enhanced MRI in detecting lymph nodes that have been invaded by tumor cells in patients with colorectal cancer. This study will be performed in addition to any ongoing routine care and will not serve as a substitute for any imaging tests that would be routinely performed prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with histologically confirmed colorectal cancer
* Planned for surgical resection of tumor

Exclusion Criteria:

* Contraindications for MRI
* Contraindication or known allergy to ferumoxytol or parental iron products (e.g. iron sucrose, iron dextran, etc.)
* Planned chemotherapy or radiation treatment prior to surgical resection of primary tumor
* Uncontrolled serious medical illness
* Unable or unwilling to give informed consent
* Pregnancy
* Breastfeeding women
* Clinically documented or known risk of primary or secondary iron overloading including history of thalassemia, sickle cell anemia, hereditary hemochromatosis or first-degree relative with known hemochromatosis, multiple transfusions for any reason within the past 5 years, or use of over-the-counter ferrous sulfate without the supervision of his/her doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Prospectively evaluate the diagnostic accuracy of ferumoxytol-enhanced MRI in the setting of colorectal cancer with histopathologic analysis as the gold standard. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Potenta, MD, PhD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States